CLINICAL TRIAL: NCT01253265
Title: Multiple-Dose, Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LY2439821 in Japanese Patients With Rheumatoid Arthritis on Concomitant Methotrexate Treatment
Brief Title: A Study in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13061; I1F-JE-RHAL (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 30 mg LY2439821 (Experimental): Administered subcutaneously at Week 0, 1, 2, 4, 6, 8 and 10
  Interventions: Drug: LY2439821
- 80 mg LY2439821 (Experimental): Administered subcutaneously at Week 0, 1, 2, 4, 6, 8 and 10
  Interventions: Drug: LY2439821
- 180 mg LY2439821 (Experimental): Administered subcutaneously at Week 0, 1, 2, 4, 6, 8 and 10
  Interventions: Drug: LY2439821
- Placebo (Placebo Comparator): Placebo is administered subcutaneously in the same manner as active drug in each dose group
  Interventions: Drug: Placebo
- 120 mg LY2439821 (Experimental): Administered subcutaneously at 240 mg as a single loading dose followed by 120 mg every week
  Interventions: Drug: LY2439821

INTERVENTIONS:
Drug: LY2439821 — Administered subcutaneously
  Arms: 120 mg LY2439821; 180 mg LY2439821; 30 mg LY2439821; 80 mg LY2439821
Drug: Placebo — Administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple doses of LY2439821 in Japanese patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory male or female patients between the ages of 20 and 75 years
* Male patients: Agree to use a reliable method of birth control during the study including barrier contraceptives or a monogamous relationship with a partner who is not child bearing. Female patients: Are women who test negative for pregnancy at the time of entry based on a pregnancy test and are not breast feeding. Women of child bearing potential must agree to use a reliable method of birth control during the study.
* Patients who are between the body weight of 40 and 105 kilogram (kg)
* Patients who have an established diagnosis of Rheumatoid Arthritis (RA)
* Patients who have C reactive protein (CRP) measurement greater than the upper limit of normal or erythrocyte sedimentation rate of at least 28 millimeters per hour (mm/hr)
* Patients who have been treated with regular use of Methotrexate (MTX) for at least 12 weeks, and stable treatment (at least 7.5 milligrams per week (mg/week)) for at least 8 weeks
* Patients who have given written informed consent approved by the Sponsor and the Institutional Review Board (IRB) governing the investigational site
* Patients who have reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Patients who use oral corticosteroids at average daily doses of >10 mg/day of prednisone or its equivalent or use of variable doses of oral corticosteroids within the last 4 weeks
* Patients who have had a live vaccination within the last 12 weeks, or intend to have a live vaccination during the course of the study, or have participated in a vaccine clinical study within the last 12 weeks
* Patients who have a diagnosis of any systemic inflammatory condition other than RA
* Patients who have evidence of active vasculitis or uveitis
* Patients who have a diagnosis of Felty's syndrome
* Patients who have had surgical treatment of a joint within the last 8 weeks, or will require it during the study
* Patients who have had lymphoma, leukemia, or any malignancy within the last 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease
* Patients who have suffered a serious bacterial infection within the last 12 weeks, or a recent or ongoing infection
* Patients who have an evidence or suspicion of active tuberculosis (TB) by medical history, physical examination, and/or chest radiograph or documentation of TB by a positive purified protein derivative (PPD) test
* Patients who have uncontrolled arterial hypertension characterized by a systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg
* Patients who have an evidence of positive hepatitis B (HBV) surface antigen, positive hepatitis B surface antibody, positive hepatitis B core antibody, or hepatitis B DNA (HBV DNA); an evidence of human immunodeficiency virus (HIV), evidence of hepatitis B; or an evidence of hepatitis C
* Patients who have clinical laboratory test results at entry that are outside the normal reference range, or results with unacceptable deviations that are considered clinically significant by the investigator
* Patients who have a serum creatinine >2.0 milligrams per deciliter (mg/dL)
* Patients who have known hypogammaglobulinemia or a serum immunoglobulin (Ig) G (IgG), IgM, or IgA concentration less than the lower limit of normal
* Patients who have an abnormality in the 12 lead electrocardiogram (ECG).
* Patients who have donated of blood more than 200 mL within the past 30 days, or more than 400 milliliters (mL) within the past 90 days
* Patients who are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an off label use of an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. For unapproved Disease-Modifying Anti-Rheumatic Drug (DMARDs), have received 30 days or 5 fold of the half life prior to inclusion whichever is longer
* Patients who previously completed or withdrawn from this study or any other study investigating LY2439821
* Patients who have been treated with any biologic DMARD currently or previously for 5 half lives
* Patients who have had serious reaction to other biologic Disease-Modifying Anti-Rheumatic Drug (DMARDs)
* Patients who have received non biologics DMARDs (other than MTX, sulfasalazine, bucillamine or hydroxychloroquine)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- Japan (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shimane
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 Milligram (mg) LY2439821; 80 mg LY2439821; 180 mg LY2439821: Administered subcutaneously at Week 0, 1, 2, 4, 6, 8 and 10
- 120 mg LY2439821: 240 mg LY2439821 was administered subcutaneously (loading dose) at Week 0, followed by 120 mg LY2439821 administered subcutaneously weekly from Week 1 through Week 10
Period: Overall Study
Arm/Group | 30 Milligram (mg) LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 5 | 6 | 6 | 6 | 7
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Met Predefined Discontinuation Criteria | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (15.4) | 56.8 (7.2) | 61.7 (11.3) | 52.5 (14.0) | 60.1 (7.7) | 57.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 3 | 4 | 5 | 22
  Male | 2 | 0 | 3 | 2 | 3 | 10
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 6 | 6 | 6 | 6 | 8 | 32
Region of Enrollment [Number; unit: participants]
  Japan | 6 | 6 | 6 | 6 | 8 | 32
C-Reactive Protein (CRP) [Median (Full Range); unit: milligrams per liter (mg/L)] | 7.950 [5.00 to 25.10] | 11.750 [2.00 to 50.10] | 3.500 [2.80 to 12.80] | 31.000 [9.30 to 95.20] | 5.650 [1.10 to 50.10] | 9.700 [1.10 to 95.20]
Erythrocyte Sedimentation Rate (ESR) [Median (Full Range); unit: millimeters per hour (mm/h)] | 28.0 [7 to 87] | 53.5 [23 to 107] | 26.0 [4 to 50] | 42.5 [22 to 81] | 25.5 [9 to 48] | 29.5 [4 to 107]
Neutrophils [Median (Full Range); unit: 10^9 cells per liter (GI/L)] | 6.763 [3.13 to 7.67] | 4.293 [2.59 to 11.12] | 3.857 [2.59 to 5.26] | 6.056 [4.63 to 7.56] | 6.757 [4.14 to 8.97] | 5.261 [2.59 to 11.12]
Lymphocytes [Median (Full Range); unit: 10^9 cells per liter (GI/L)] | 0.993 [0.42 to 2.62] | 1.156 [0.69 to 2.19] | 1.187 [0.88 to 2.01] | 1.379 [0.67 to 2.45] | 1.295 [1.06 to 2.29] | 1.275 [0.42 to 2.62]
Duration of Rheumatoid Arthritis (RA) [Mean (Standard Deviation); unit: years] | 10.9 (11.8) | 7.9 (9.7) | 6.8 (12.0) | 5.6 (4.1) | 3.6 (3.2) | 6.8 (8.5)
Weekly dose of Methotrexate (MTX) [Mean (Standard Deviation); unit: milligrams per week (mg/wk)] | 8.33 (0.82) | 8.33 (0.82) | 8.00 (0.00) | 9.00 (1.10) | 9.06 (1.66) | 8.58 (1.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Clinically significant events were defined as serious and other non-serious adverse events. A summary of serious and all other non-serious adverse events is located in the Reported Adverse Event module.
Time Frame: Baseline up to 26 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0
  Other Adverse Events | 4 | 5 | 3 | 3 | 6

2. Secondary Outcome: Percentage Change From Baseline to 16 Week Endpoint in C-Reactive Protein
Description: C-reactive protein (CRP) is a disease related biomarker and measured in milligrams per liter.
Time Frame: Baseline, 16 weeks
Population: All randomized participants.
Measure: Median (Full Range); unit: percentage change in C-Reactive Protein
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage change in C-Reactive Protein | -88.75 [-98.6 to -66.7] | -73.81 [-98.8 to 180.0] | -17.04 [-48.4 to 150.0] | -95.47 [-99.3 to 100.0] | -8.07 [-82.8 to 186.2]

3. Secondary Outcome: Percentage Change From Baseline to 16 Week Endpoint in Erythrocyte Sedimentation Rate (ESR)
Description: Erythrocyte Sedimentation Rate (ESR) is a disease related biomarker and measured in millimeters per hour (mm/h).
Time Frame: Baseline, 16 weeks
Population: All randomized participants.
Measure: Median (Full Range); unit: percentage change in ESR
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
percentage change in ESR | -44.50 [-80.0 to -16.7] | -35.05 [-76.1 to 13.3] | -3.75 [-37.9 to 100.0] | -73.08 [-92.7 to -5.6] | -12.62 [-54.5 to 137.5]

4. Secondary Outcome: Change From Baseline to 26 Week Endpoint in Neutrophil Counts
Time Frame: Baseline, 26 weeks
Population: All randomized participants.
Measure: Median (Full Range); unit: 10^9 cells per liter (GI/L)
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
10^9 cells per liter (GI/L) | 0.681 [-5.77 to 5.84] | -0.559 [-2.62 to 5.62] | -0.170 [-0.87 to 2.72] | -2.677 [-2.87 to -0.70] | -0.641 [-2.94 to 2.29]

5. Secondary Outcome: Change From Baseline to 26 Week Endpoint in Lymphocyte Counts
Time Frame: Baseline, 26 weeks
Population: All randomized participants.
Measure: Median (Full Range); unit: 10^9 cells per liter (GI/L)
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
10^9 cells per liter (GI/L) | 0.189 [-1.19 to 1.23] | -0.011 [-0.54 to 1.25] | -0.184 [-0.37 to 0.09] | 0.138 [-0.15 to 0.65] | 0.085 [-0.56 to 0.24]

6. Secondary Outcome: Pharmacokinetics - Area Under the Concentration-time Curve (AUC) at Steady State (ss)
Description: AUCτ,ss= area under the concentration versus time curve (τ) at steady state (ss)
Time Frame: Week 10 pre-dose up to 2 weeks post-dose (Week 12)
Population: All randomized participants with analyzable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms•day per milliliter(μg•day/mL)
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821
Number analyzed (Participants) | 5 | 6 | 6 | 6
micrograms•day per milliliter(μg•day/mL) | 77.2 (26) | 151 (44) | 437 (42) | 208 (48)

7. Secondary Outcome: Pharmacokinetics - Maximum Plasma Drug Concentration (Cmax) at Steady State (ss)
Description: Cmax,ss = maximum observed drug concentration (Cmax) at steady state (ss)
Time Frame: Week 10 pre-dose up to 2 weeks post-dose (Week 12)
Population: All randomized participants with analyzable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821
Number analyzed (Participants) | 5 | 6 | 6 | 6
micrograms per milliliter (μg/mL) | 7.05 (26) | 13.5 (43) | 39.3 (42) | 33.1 (56)

8. Secondary Outcome: Pharmacokinetics - Time of Maximum Observed Drug Concentration (Tmax) at Steady State (ss)
Description: tmax,ss = time of maximum observed drug concentration (tmax) at steady state (ss)
Time Frame: Week 10 pre-dose up to 2 weeks post-dose (Week 12)
Population: All randomized participants with analyzable pharmacokinetic data.
Measure: Median (Full Range); unit: days
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821
Number analyzed (Participants) | 5 | 6 | 6 | 6
days | 1.96 [1.91 to 7.00] | 1.93 [1.89 to 3.97] | 1.95 [1.88 to 2.02] | 3.89 [1.93 to 3.99]

ADVERSE EVENTS:
Arm/Group | 30 mg LY2439821 | 80 mg LY2439821 | 180 mg LY2439821 | 120 mg LY2439821 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 3/6 | 3/6 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 30 mg LY2439821 (N=6) | 80 mg LY2439821 (N=6) | 180 mg LY2439821 (N=6) | 120 mg LY2439821 (N=6) | Placebo (N=8)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Administration site reaction (General disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (3) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menopausal symptoms (Reproductive system and breast disorders) | 1/4 (1) | 0 (0) | 0/3 (0) | 0/4 (0) | 0/5 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days